CLINICAL TRIAL: NCT00612014
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-ranging Study to Assess the Efficacy and Safety of TZP-101 When Administered as a 30 Minute I.V. Infusion to Subjects With Severe Gastroparesis Due to Diabetes Mellitus
Brief Title: Safety and Efficacy of IV Infusion of Investigational Agent (TZP-101) in Patients With Severe Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZP-101-CL-G004; 2007-003279-38
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: delayed gastric emptying; symptomatic gastroparesis; diabetes mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Glucose; Water; ulimorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Placebo Comparator)
  Interventions: Drug: 5% dextrose in water
- 2 (Experimental): 40 micrograms/kg
  Interventions: Drug: TZP-101
- 3 (Experimental): 80 micrograms/kg
  Interventions: Drug: TZP-101
- 4 (Experimental): 160 micrograms/kg
  Interventions: Drug: TZP-101
- 5 (Experimental): 320 microgram/kg
  Interventions: Drug: TZP-101
- 6 (Experimental): 600 microgram/kg
  Interventions: Drug: TZP-101

INTERVENTIONS:
Drug: 5% dextrose in water — 60 ml IV infusion over 30 minutes
  Other Names: D5W
  Arms: 1
Drug: TZP-101 — 40 micrograms/kg iv 2ml/minute for 30 minutes
  1 infusion/day for 4 consecutive days
  Arms: 2
Drug: TZP-101 — 80 micrograms/kg iv 2ml/minute for 30 minutes
  1 infusion/day for 4 consecutive days
  Arms: 3
Drug: TZP-101 — 160 micrograms/kg iv 2ml/minute for 30 minutes
  1 infusion/day for 4 consecutive days
  Arms: 4
Drug: TZP-101 — 320 micrograms/kg iv 2ml/minute for 30 minutes
  1 infusion/day for 4 consecutive days
  Arms: 5
Drug: TZP-101 — 600 micrograms/kg iv 2ml/minute for 30 minutes
  1 infusion/day for 4 consecutive days
  Arms: 6

SUMMARY:
The purpose of this study is to determine whether TZP-101 is effective in the treatment of symptomatic gastroparesis due to diabetes.

DETAILED DESCRIPTION:
Subjects are randomized according to an adaptive randomization procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject has type 1 or type 2 diabetes mellitus
* Subject has documented diagnosis of gastroparesis (all of the following apply):

  * Confirmed delayed gastric emptying (see Appendix IV; properly conducted gastric emptying assessments within last 6 months acceptable)
  * AND a minimum 3 month history of relevant symptoms for gastroparesis (chronic postprandial fullness, bloating, epigastric discomfort, early satiety, belching after meal, postprandial nausea, vomiting).
  * AND a mean Gastroparesis Cardinal Symptom Index (GCSI) Score (2 week recall version) of ≥ 2.66
  * AND it is confirmed by endoscope that there are no obstructive lesions in the esophagus or stomach (endoscopy within prior 3 months acceptable)
* Subject has never had a gastrectomy, nor major abdominal surgery or any evidence of bowel obstruction within the previous 12 months
* Dosage of any concomitant medications has been stable for at least 3 weeks
* HbA1c level is ≤ 10.0%
* Subject has a BMI < 30
* Subject body weight is ≤ 100 kg
* If female, post-menopausal for the past 12 months, surgically sterile (i.e. tubal ligation, hysterectomy), or using an adequate method of birth control (i.e., oral contraceptives, double barrier method, IUD cover) or sterilized partner

Exclusion Criteria:

* Subject has acute severe gastroenteritis
* Subject has a gastric pacemaker
* Subject is on chronic parenteral feeding
* Subject has daily persistent severe vomiting
* Subject has pronounced dehydration
* Subject has had diabetic ketoacidosis in last 4 weeks
* Subject has a history of eating disorders (anorexia nervosa, binge eating, bulimia)
* Subject has a marked baseline prolongation of QT/QTc interval (repeated demonstration of a QTc interval >450 ms for male / >470 ms for female)
* Subject has a history of additional risk factors for Torsades de Pointes (heart failure, chronic hypokalemia, family history of Long QT Syndrome)
* Subject requires use of concomitant medication that prolongs the QT interval

  * List provided to clinical sites
* Subject has history of cardiovascular ischemia in previous 12 months or acute myocardial infarction (MI) or unstable angina
* Subject requires use of concomitant medication that is known to interact with isoenzyme CYP3A4 and the combination with an CYP3A4 inhibitor is known to introduce a clinically significant drug interaction

  * List provided to clinical sites
* Subject has a history of psychiatric disorder or cognitive impairment that would interfere with participation in the study
* Subject has a history of alcoholism
* Subject is taking regular daily narcotics
* Subject has a known history of Hep B, Hep C or HIV
* Subject has severely impaired renal function (creatinine clearance < 30 mL/min)
* Subject has severe impairment of liver function, defined as albumin level ≤ 2.5 gm/dL and/or prothrombin time >6 seconds over control (INR > 2.3)
* Subject has participated in an investigational study within 30 days prior to or received TZP-101 within 90 days prior to study initiation
* Subject is pregnant or is breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean Gastroparesis Cardinal Symptom Index score (24 hour recall version) across the four days of dosing. Baseline is the average of the scores collected across the 4 days just prior to admission for dosing. | after 4 dosing days

SECONDARY OUTCOMES:
Cumulative GSA score after each dosing event and after all dosing events | every 30 minutes for 4 hours

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - California Pacific Medical Center, San Francisco, California
  - Central Indiana Gastroenterology Group, Anderson, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
- Aarhus University Hospital, Aarhus, Denmark
- Amrita Institute of Medical Sciences Research Center (AIMS), Kochi, Kerala, India
- Haukeland University Hospital, Bergen, Norway
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Manchester Royal Infirmary, Manchester
  - Royal Hallamshire Hospital, Sheffield